CLINICAL TRIAL: NCT06286631
Title: Quantitative Rating Scale Based on Preoperative Prediction of Lymph Node Dissection in Patients With Thyroid Cancer
Brief Title: Prediction of Lymph Node Metastasis in Patients With Thyroid Malignancy by a New Scale
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: Rating scale-202402
Record Dates: First submitted 2024-02-07; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Papillary Thyroid Cancer
Keywords: Papillary Thyroid Cancer; pre-operative; Prophylactic lymph node dissection; lymphatic node transfer; Multi-factor data
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Past Medical Records Group: Sample size:500 Whether control group:No Name of exposure factor:papillary thyroid cancer Exposure factor type:Other Description of exposure factor:None
- Clinical Validation Group: Sample size:300 Whether control group:No Name of exposure factor:papillary thyroid cancer Exposure factor type:Other Description of exposure factor:None

SUMMARY:
The incidence of papillary thyroid cancer (PTC) has been on the rise in recent years, and 20%-50% of PTC patients will have lymph node metastasis. Lymph node involvement in PTC patients is usually related to the recurrence of PTC after surgery, and 30% of patients recur without lymph node dissection, with the risk of central cervical lymph node metastasis being the greatest, so it seems to be a good choice to perform lymph node dissection on patients after thyroidectomy, but in fact, there are controversies at home and abroad as to whether to perform lymph node dissection or not. The 2021 Chinese Society of Clinical Oncology (CSCO) guidelines for the diagnosis and treatment of differentiated thyroid cancer state that prophylactic central lymph node dissection (PCND) may increase the incidence of postoperative complications, but due to the high metastatic rate of PTC and the ability of PCND to effectively prevent recurrence and reoperation, countries in the East Asian region perform prophylactic lymph node dissection on almost all patients with PTC. However, for more countries in Europe and the United States, performing PCND has become a non-essential, individualized option. The aim of this study is to collect multifactorial data from more than 1,000 patients who have undergone previous thyroidectomy from 2021 to 2023, and to develop a novel scoring scale that can be used to individualize patients' scores based on a variety of factors prior to surgery, so that patients can be more accurately predicted to have lymph node metastasis and need prophylactic lymph node dissection prior to surgery, and patients who do not need dissection can avoid surgery. For patients who do not need lymph node dissection, complications caused by surgery can be avoided, while for patients who do have lymph node metastasis, recurrence of their cancer can be prevented. This will change the status quo of not being able to accurately determine the actual situation through simple preoperative examination or performing prophylactic lymph node dissection for all PTC patients.

DETAILED DESCRIPTION:
1. Patient characteristics: the inclusion criteria were as follows:1. patients with papillary thyroid cancer;2. minimum age of 16 years old and maximum age of 80 years old. Exclusion criteria:1. age less than 16 years old;2. postoperative pathology suggesting that there are other types of tumors, such as medullary carcinoma or undifferentiated carcinoma. 2,.Data collection: Investigators collected multifactorial data on about 1000 patients who had undergone previous thyroidectomy from 2021-2023, including gender, height, age, weight, BMI, diameter of the tumor in the primary focus, tumor limitation in the primary focus, lymph node metastasis, and tumor invasion, preoperative ultrasonographic manifestations, preoperative laboratory results, pathological results, and genetic testing results. From these, the available data were screened and retained for analysis. 3.Data analysis: According to the retained data after screening, classical machine learning algorithms will be used for feature selection to select the factors with greater correlation with the results, and then with the help of data visualization, the specific quantitative relationship between each factor and the results will be determined according to the distribution of the available data, and the quantitative scoring table will be created. 4. Clinical validation: The completed quantitative rating scale investigators will be validated in the clinic. Investigators will use the scale to score new patients to assess whether participants need prophylactic lymph node dissection, and then evaluate the accuracy of the quantitative scale according to the intraoperative or postoperative situation.

ELIGIBILITY:
Inclusion Criteria:

* Papillary thyroid cancer
* Conscious and able to communicate normally
* Age 16-80 years

Exclusion Criteria:

* Preoperative or postoperative pathology suggests other types of tumors, such as medullary carcinoma or undifferentiated carcinoma.
* Less than 16 years of age

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From 2021 to 2023, 500 patients with previous papillary thyroid cancer surgery were selected at the Second Affiliated Hospital of Xi'an Jiaotong University for the quantitative rating scale, as well as 300 newly admitted papillary thyroid cancer patients for subsequent validation.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Height | up to three years
  The height indicator will summarize the data in "meters".
Weight | up to three years
  The weight indicator will summarize data in "kilograms".
Age | up to three years
  Age will be aggregated using "years" as the unit of measurement.
Genders | up to three years
  Data will be summarized in terms of "male" and "female" as units of measurement.
BMI | up to three years
  BMI will be summarized in "kg/m^2".
Whether lymph node dissection was performed during previous surgery | up to three years
  Data will be summarized using "yes" or "no" for whether lymph node dissection was performed during previous surgery.
Tumor Diameter Size | up to three years
  Tumor diameter size will be summarized in "millimeters".
Tumor limitation of the primary focus | up to three years
  Tumor limitation of primary foci will be summarized using "single/multiple" and "unilateral/bilateral".
Extratumoral invasion | up to three years
  Extra-tumor focal invasion will be summarized with a "yes" or "no" to the data.
Pathologic lymph node metastasis | up to three years
  Pathological lymph node metastases will be summarized with "yes" or "no" data.
Tumor cystic solidity on preoperative ultrasound | up to three years
  Pre-operative ultrasound tumor cysticity will be summarized as "cystic" or "solid".
Preoperative ultrasound tumor echo intensity | up to three years
  Preoperative ultrasound tumor echo intensity will be summarized as "high echo" or "moderate echo" or "low echo" or "very low echo".
Preoperative ultrasound tumor boundaries | up to three years
  Preoperative ultrasound tumor boundaries will be summarized as "clear" or "unclear".
Preoperative ultrasound tumor for the presence of calcifications | up to three years
  Preoperative ultrasound tumors will be summarized with "yes" or "no" for the presence of calcifications.
Preoperative ultrasound tumor aspect ratios | up to three years
  Preoperative ultrasound tumor aspect ratios will be summarized with ">1" or "<1" data
Preoperative ultrasound for enlarged cervical lymph nodes | up to three years
  Preoperative ultrasound of cervical lymph nodes for enlargement will be summarized as "yes" or "no".
TSH | up to three years
  The TSH indicator will summarize data in "mlU/L".
TPOAb | up to three years
  The TPOAb indicator will summarize data in "lU/mL".
TgAb | up to three years
  The TgAb indicator will summarize data in "lU/mL".
Calcium | up to three years
  The Calcium indicator will summarize data in "mmol/L".
B-raf gene mutation | up to three years
  B-raf mutations will be summarized as "wild type" or "mutant".

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

DOCUMENTS (2):
  • Study Protocol (2023-10-29): https://cdn.clinicaltrials.gov/large-docs/31/NCT06286631/Prot_000.pdf
  • Informed Consent Form (2023-10-29): https://cdn.clinicaltrials.gov/large-docs/31/NCT06286631/ICF_001.pdf